CLINICAL TRIAL: NCT02567227
Title: Cognitive Intervention to Improve Simple and Complex Walking
Brief Title: Cognitive Remediation to Improve Mobility in Sedentary Seniors
Acronym: CREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-4752; R01AG050448-01 (NIH)
Record Dates: First submitted 2015-08-17; First posted 2015-10-02 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Mobility Limitation; Motor Activity; Difficulty Walking; Cognitive Ability General
MeSH Terms: conditions — Mobility Limitation; Motor Activity | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Remediation (Experimental): An individualized computerized cognitive remediation program.
  Interventions: Other: Cognitive Remediation
- Active control (Active Comparator): Individualized computer based exposure and interactive health education classes.
  Interventions: Other: Active Control

INTERVENTIONS:
Other: Cognitive Remediation — This computerized program has successfully been used by seniors in different settings. It trains a number of cognitive processes including attention and Executive Function.The Cognitive Remediation (CREM) training is constructed based on the program's built in baseline cognitive evaluation.
  Arms: Cognitive Remediation
Other: Active Control — Computer, multimedia and group based health education programs.
  Arms: Active control

SUMMARY:
The investigators propose to conduct a single-blind randomized clinical trial to test the efficacy of a computerized cognitive remediation intervention program on improving locomotion in sedentary seniors, a group at an especially high risk for disability. The hypothesis is that executive functions will respond to the cognitive remediation program and in turn enhance locomotion.

DETAILED DESCRIPTION:
Emerging evidence indicates that Executive Functions play an important role in maintaining locomotion in aging and preventing mobility disabilities. However, use of cognitive training programs to improve executive functions as a strategy to increase mobility has not been explored. Exciting results from the preliminary study support the efficacy and feasibility of the cognitive remediation approach to improve locomotion in older adults.

The premise of this clinical trial is that disability among seniors is a potentially preventable chronic condition rather than an irreversible consequence of aging and disease. The investigators proposed novel approach to locomotion has the potential to shift treatment paradigms in the field of disability by introducing cognitive approaches to mobility that can be applied to prevention and rehabilitation in diverse settings. Through this 'proof of concept' secondary prevention trial the investigators will fill an important gap in knowledge for practicing evidence-based medicine and developing effective interventions for a major health outcome affecting a substantial proportion of the U.S. aging population.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 70 and older, residing in the community.
2. Plan to be in area for next year.
3. Able to speak English at a level sufficient to undergo our cognitive assessment battery.
4. Ambulatory. Subjects are classified as 'non-ambulatory' if they are unable to leave the confines of their home and attend a clinic visit.
5. Gait velocity ≤1 m/s.
6. Short Physical Performance Battery score ≤9.

Exclusion Criteria:

1. Presence of dementia identified by any one of the following: Telephone based Memory Impairment Screen score (T-MIS) of <5, Alzheimer's Disease 8 (AD8) ≥ 2. Or dementia diagnosed by baseline cognitive assessment.
2. Serious chronic or acute illness such as cancer (late stage, metastatic, or on active treatment), chronic pulmonary disease on ventilator or continuous oxygen therapy or active liver disease.
3. Mobility limitations solely due to musculoskeletal limitation or pain (e.g., severe osteoarthritis) that prevent subjects from completing mobility tests. Presence of arthritis will not be used to exclude subjects if they can complete the mobility tasks.
4. Any medical condition or chronic medication use (e.g., neuroleptics) that will compromise safety or affect cognitive functioning or terminal illness with life expectancy less than 12 months.
5. Presence of progressive, degenerative neurologic disease (e.g., Parkinson's disease or ALS).
6. Hospitalized in the past 6 months for severe illness or surgery that specifically affects mobility (e.g. hip or knee replacement) and that prevent subjects from completing mobility tests or plans for surgery affecting mobility in the next 6 months.
7. Severe auditory or visual loss.
8. Active psychoses or psychiatric symptoms (such as agitation) noted during the clinic visit that will prevent completion of study protocols.
9. Living in nursing home.
10. Participation in other intervention trial or observational studies. -

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 383 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Verghese, MD, Principal Investigator — Albert Einstein College of Medicine; Roee Holtzer, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Result] Verghese J, Mahoney J, Ambrose AF, Wang C, Holtzer R. Effect of cognitive remediation on gait in sedentary seniors. J Gerontol A Biol Sci Med Sci. 2010 Dec;65(12):1338-43. doi: 10.1093/gerona/glq127. Epub 2010 Jul 19. PMID 20643703
- [Derived] Verghese J, Mahoney JR, Ayers E, Ambrose A, Wang C, Holtzer R. Computerised cognitive remediation to enhance mobility in older adults: a single-blind, single-centre, randomised trial. Lancet Healthy Longev. 2021 Sep;2(9):e571-e579. doi: 10.1016/s2666-7568(21)00173-2. Epub 2021 Sep 2. PMID 34522910
- [Derived] Verghese J, Ayers E, Mahoney JR, Ambrose A, Wang C, Holtzer R. Cognitive remediation to enhance mobility in older adults: the CREM study. Neurodegener Dis Manag. 2016 Dec;6(6):457-466. doi: 10.2217/nmt-2016-0034. Epub 2016 Nov 4. PMID 27813452

RESULTS

PARTICIPANT FLOW:
Period: 9 Weeks
Arm/Group | Cognitive Remediation | Active Control
Started | 192 | 191
Completed | 158 | 167
Not Completed | 34 | 24
Not completed — Adverse Event | 5 | 5
Not completed — Withdrawal by Subject | 18 | 8
Not completed — Study suspended due to COVID-19 pandemic | 11 | 11
Period: 6 Month
Arm/Group | Cognitive Remediation | Active Control
Started | 158 | 167
Completed | 113 | 127
Not Completed | 45 | 40
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 43 | 40
Period: 12 Months
Arm/Group | Cognitive Remediation | Active Control
Started | 113 | 127
Completed | 82 | 93
Not Completed | 31 | 34
Not completed — Lost to Follow-up | 31 | 32
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: Includes all participants who were randomized. Excludes participants diagnosed with dementia post-hoc (n=6 in Experimental; n=5 in Active Comparator)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Remediation | Active Control | Total
Number analyzed (Participants) | 186 | 186 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.94 (5.66) | 77.18 (5.61) | 77.03 (5.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 136 | 271
  Male | 51 | 50 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 34 | 62
  Not Hispanic or Latino | 151 | 142 | 293
  Unknown or Not Reported | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 93 | 90 | 183
  White | 57 | 47 | 104
  More than one race | 28 | 34 | 62
  Unknown or Not Reported | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 186 | 186 | 372
Gait Speed, cm/s [Mean (Standard Deviation); unit: centimeters per second] — Gait speed during normal walking.
  centimeters per second | 75.82 (17.73) | 75.92 (16.81) | 75.87 (17.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Speed During Single and Dual-task Conditions.
Description: Between group difference in change per arm of gait speed (centimeters/second) measured during normal pace walking and walking while talking conditions using an instrumented walkway (GAITRite® electronic walkway system).
Time Frame: Baseline and 2 months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: centimeters per second
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
centimeters per second
  Normal pace walking | 1.73 (0.94) | 2.76 (0.91)
  Walking while talking | 6.02 (1.16) | 5.43 (1.13)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (Mild Cognitive Impairment (MCI) or cognitively normal) were used to compare changes in speed during normal pace walking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -1.03, 95% CI 2-sided [-3.60 to 1.54], Standard Error of Mean 1.30 — Estimates with standard errors are from linear mixed effect models adjusted for age, sex, education years, comorbidities, pain, cardiac fitness, and cognitive status
Statistical Analysis 2: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in speed during walking while talking pre and post intervention; Test type: Superiority; P-values from linear mixed effects models adjusted for age, sex, education years, comorbidities, pain, cardiac fitness, and cognitive status; Mean Difference (Net) = 0.59, 95% CI 2-sided [-2.59 to 3.76], Standard Error of Mean 1.61 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Short Physical Performance Battery (SPPB).
Description: Between group difference in change per arm in mobility measured using the SPPB. The SPPB is comprised of balance, chair rise, and gait speed tests. A score is assigned in each of these three areas (0-4), and summed to obtain an overall summary score (0-12, higher better).
Time Frame: Baseline and 2 months
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
score on a scale | 0.70 (0.13) | 0.85 (0.12)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in SPPB scores pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.49 to 0.20], Standard Error of Mean 0.17 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Stride Length.
Description: Between group difference in change per arm in stride length (cm) collected during normal walking and walking while talking conditions on an instrumented walkway.
Time Frame: Baseline and 2 months
Population: Includes all participants who were randomized. Excludes participants diagnosed with dementia post-hoc (n=6 Experimental; n=5 Active Comparator).
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
centimeters
  Walking while talking stride length | 3.09 (1.08) | 2.26 (1.05)
  Normal walking stride length | 0.13 (0.81) | 2.08 (0.66)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in stride length during walking while talking pre and post intervention; Test type: Superiority; Mean Difference (Net) = 0.83, 95% CI 2-sided [-2.13 to 3.79], Standard Error of Mean 1.50 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cognitive Remediation vs Active Control; Unadjusted linear mixed effects models were used to compare changes in stride length during normal walking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -1.95, Standard Error of Mean 1.04 — Estimates with standard errors are from linear mixed effect models

4. Secondary Outcome: Gait Variability.
Description: Between group difference in change per arm in gait stride length variability, measured in standard deviation units, collected during normal walking and walking while talking on an instrumented walkway. Gait variability is defined as differences in length from one stride to the next.
Time Frame: Baseline and 2 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: standard deviation
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
standard deviation
  Normal walking gait variability | -0.37 (0.25) | -0.13 (0.24)
  Walking while talking gait variability | -0.52 (0.26) | -0.08 (0.26)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in stride length variability during normal walking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.91 to 0.43], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in stride length variability during walking while talking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.44, 95% CI 2-sided [-1.16 to 0.27], Standard Error of Mean 0.36 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Variability in Gait Domains
Description: Between group difference in change per arm in gait domains (summary measures reported as standard deviation units) derived from factor analysis of quantitative gait variables collected on an instrumented walkway during normal walking and walking while talking. Based on previous findings of gait patterns, pace, rhythm and variation factors are defined (using z-scores based on mean and standard deviation at baseline). Higher values are indicative of better performance for pace and rhythm factors and indicative of worse performance for variation factors.
Time Frame: Baseline and 2 Months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: standard deviation
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
standard deviation
  Normal walking pace | 0.21 (0.14) | 0.37 (0.11)
  Normal walking rhythm | 0.36 (0.12) | 0.25 (0.10)
  Normal walking variation | 0.07 (0.16) | -0.15 (0.13)
  Walking while talking pace | 0.75 (0.15) | 0.60 (0.15)
  Walking while talking rhythm | 0.72 (0.15) | 0.74 (0.19)
  Walking while talking variation | -0.24 (0.11) | -0.22 (0.15)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the pace domain during normal pace walking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.51 to 0.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the rhythm domain during normal pace walking pre and post intervention; Test type: Superiority; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.20 to 0.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the variation domain during normal pace walking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.53 to 0.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the pace domain during walking while talking pre and post intervention; Test type: Superiority; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.27 to 0.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the rhythm domain during walking while talking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.48 to 0.45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the variation domain during walking while talking pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.40 to 0.35] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Substantial Gait Speed Change.
Description: Substantial gait speed improvement is defined as change of ≥1 standard deviation units from baseline performance in gait speed measured during normal walking and walking while talking conditions.
Time Frame: Baseline and 2 Months
Population: Includes all participants who were randomized. Excludes participants diagnosed with dementia post-hoc (n=6 Experimental; n=5 Active Comparator) and participants who did not complete the 2 month follow-up assessment (n=34 Experimental; n=24 Active Comparator).
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 152 | 162
Participants
  Substantial normal walking speed improvement: Improved walking speed ≥1 standard deviation units from baseline | 10 | 11
  Substantial normal walking speed improvement: Did not improve walking speed ≥1 standard deviation units from baseline | 142 | 151
  Substantial walking while talking speed improvement: Improved walking speed ≥1 standard deviation units from baseline | 23 | 25
  Substantial walking while talking speed improvement: Did not improve walking speed ≥1 standard deviation units from baseline | 129 | 137
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Logistic model for treatment effect on substantial improvement in normal velocity adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal); Test type: Superiority; Odds Ratio (OR) = 0.925, 95% CI 2-sided [0.369 to 2.319]
Statistical Analysis 2: Comparison: Cognitive Remediation vs Active Control; Logistic model for treatment effect on substantial improvement in walking while talking velocity adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal); Test type: Superiority; Odds Ratio (OR) = 0.961, 95% CI 2-sided [0.516 to 1.789]

7. Secondary Outcome: Flanker Task.
Description: Between group difference in change per arm on the Flanker task, a measure of speed of processing, attention and inhibitory control. Scoring is based on reaction time in milliseconds (ms) and calculated as the difference in reaction time that it takes a person, on average, to respond to an incongruent minus congruent stimulus. Lower values reflect better outcome.
Time Frame: Baseline and 2 Months
Population: Includes all participants who were randomized. Excludes participants diagnosed with dementia post-hoc (n=6 Experimental; n=5 Active Comparator) and 86 participants (n=43 Experimental; n=43 Active Comparator) with performance inaccuracy >75%.
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 143 | 143
milliseconds | -9.05 (9.48) | -1.54 (10.55)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in Flanker performance (milliseconds) pre and post intervention; Test type: Superiority; Mean Difference (Net) = -7.52, 95% CI 2-sided [-35.45 to 20.41], Standard Error of Mean 14.17 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Digit Symbol Substitution Test.
Description: Between group difference in change per arm on the Digit Symbol Substitution Test (a subtest of the Wechsler Adult Intelligence Scale - Revised), a measure of attention, transcription and speed of processing. Scoring is based on the total number of correct responses generated during a 90-sec time interval. Scores range from 0-133 with higher scores indicating better performance.
Time Frame: Baseline and 2 Months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
score on a scale | 2.22 (0.48) | 1.21 (0.46)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes on the Digit Symbol Substitution Test pre and post intervention; Test type: Superiority; Mean Difference (Net) = 1.01, 95% CI 2-sided [-0.30 to 2.31], Standard Error of Mean 0.66 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Trail Making Test Form A.
Description: Between group difference in change per arm on Trail Making Test form A, a timed measure of attention. Scoring is based on the time required to complete the task and on accuracy. Scores range from 0-300 seconds with longer time indicating worse performance. Scores were log transformed prior to analysis.
Time Frame: Baseline and 2 Months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: log (scores on a scale)
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
log (scores on a scale) | -0.06 (0.02) | -0.07 (0.02)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Unadjusted linear mixed effects model was used to compare performance on Trail Making Test form A pre and post intervention; Test type: Superiority; Mean Difference (Net) = 0.00, Standard Error of Mean 0.03 — Estimates with standard errors are from unadjusted linear mixed effect models

10. Secondary Outcome: Trail Making Test Form B.
Description: Between group difference in change per arm on Trail Making Test form B, a timed measure of attention, set shifting and processing speed. Scoring is based on the time required to complete the task and on accuracy. Scores range from 0-300 seconds with longer time indicating worse performance. Scores were log transformed prior to analysis.
Time Frame: Baseline and 2 Months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: log (scores on a scale)
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
log (scores on a scale) | -0.10 (0.024) | -0.10 (0.02)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in performance on Trail Making Test form B pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.07 to 0.06], Standard Error of Mean 0.03 — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Controlled Oral Word Association Test.
Description: Between group difference in change per arm on the Controlled Oral Word Association Test, a verbal fluency test that measures word generation performance under specified timed phonemic and semantic conditions. Performance measured by the total number of correct words as well as the number of errors. Scores range from 25-41 seconds with higher scores indicating better performance.
Time Frame: Baseline and 2 Months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
score on a scale | 1.20 (0.56) | 0.53 (0.54)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes performance on the Controlled Oral Word Association Test pre and post intervention; Test type: Superiority; Mean Difference (Net) = 0.67, 95% CI 2-sided [-0.86 to 2.20], Standard Error of Mean 0.78 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status.
Description: Between group difference in change on the Repeatable Battery for the Assessment of Neuropsychological Status, a relatively brief battery that assesses overall level of cognitive function This battery consists of 10 neurocognitive tests measuring memory (immediate and delayed), attention, language, visuospatial abilities and executive functions. Performance is converted to standardized scores derived from a normative sample.
Time Frame: Baseline and 2 Months
Population: No outcome measure data was collected for this outcome.
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Neuroplasticity.
Description: Changes in prefrontal activation measure using functional near infra-red spectroscopy.
Time Frame: Baseline and 2 Months
Population: No outcome measure data was collected for this outcome.
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Durability
Description: Between group difference in change per arm in gait speed during normal pace and walking while talking conditions measured at six months.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: centimeters per second
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
centimeters per second
  Normal Walking Gait Speed | -0.47 (1.03) | -1.60 (0.97)
  Walking While Talking Gait Speed | 3.16 (1.30) | 1.77 (1.23)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in gait speed during normal walking pre and 6 months post intervention; Test type: Superiority; Mean Difference (Net) = 1.13, 95% CI 2-sided [-1.65 to 3.91], Standard Error of Mean 1.42 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in gait speed during walking while talking pre and 6 months post intervention; Test type: Superiority; Mean Difference (Net) = 1.40, 95% CI 2-sided [-2.12 to 4.91], Standard Error of Mean 1.79 — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Stair Climbing Time.
Description: Between group difference in change per arm in mobility and balance assessed during stair climbing, which provides a valid assessment tool for predicting disability. Scores are measured as time in seconds to climb 3 stairs with longer time indicating worse performance. Scores were log transformed prior to analysis.
Time Frame: Baseline and 2 Months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: log (seconds)
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
log (seconds) | -0.02 (0.03) | 0.01 (0.02)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Unadjusted linear mixed effects model was used to compare changes in stair climbing time pre and post intervention; Test type: Superiority; Mean Difference (Net) = -0.03, Standard Error of Mean 0.04 — Estimates with standard errors are from unadjusted linear mixed effect models

16. Secondary Outcome: Disability Scale.
Description: Between group difference in change per arm in mobility assessed by activities of daily living tasks on the Activities of Daily Living-Prevention Instrument. Scores range from 0-45 and higher scores indicate poorer function.
Time Frame: Baseline and 2 Months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
score on a scale | -0.18 (0.21) | -0.21 (0.24)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Unadjusted linear mixed effects model was used to compare changes in activities of daily living pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = 0.03, Standard Error of Mean 0.32 — Estimates with standard errors are from unadjusted linear mixed effect models

17. Other Pre Specified Outcome: The Geriatric Depression Scale (GDS).
Description: Between group difference in change per arm in depressive symptoms assessed using the 30 item GDS, scores range from 0 (not depressed) to 30 (depressed).
Time Frame: Baseline and 2 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
score on a scale | 0.41 (0.26) | 0.15 (0.21)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in depressive symptoms measured using the GDS pre and post intervention; Test type: Superiority; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.40 to 0.93], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 1]

18. Other Pre Specified Outcome: Rosenberg Self-Esteem Scale.
Description: Between group difference in change per arm in self-esteem assessed using a ten-item Likert-type scale (higher scores are better).
Time Frame: Baseline and 2 months
Population: Only baseline data was collected on this outcome measure, therefore no data was analyzed.
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 0 | 0

19. Other Pre Specified Outcome: Falls Efficacy Scale.
Description: Between group difference in change per arm in self-efficacy scores (range 0-100). Higher scores indicate less confidence.
Time Frame: Baseline and 2 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
score on a scale | 0.79 (0.69) | 0.40 (0.58)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in reported fear of falling measured on the Falls Efficacy Scale pre and post intervention; Test type: Superiority; Mean Difference (Net) = 0.39, 95% CI 2-sided [-1.38 to 2.16], Standard Error of Mean 0.90 — [estimate comment as in outcome 1, analysis 1]

20. Other Pre Specified Outcome: 12-Item Short Form Health Survey (SF-12).
Description: Between group difference in change per arm in perceptions of health and quality of life in domains that include social, physical, emotional and mental functions. The SF-12 has 12 items; two component scores capturing perceptions of mental and physical function can be derived. The Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) scores are calculated using 12 questions with a range of 0-100 (zero indicating the poorest level of health measured and 100 indicating the highest).
Time Frame: Baseline and 2 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Remediation | Active Control
Number analyzed (Participants) | 186 | 186
score on a scale
  Physical Component Summary | 0.31 (0.45) | 0.52 (0.45)
  Mental Component Summary | -0.76 (0.50) | -1.17 (0.53)
Statistical Analysis 1: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the physical health score of the SF-12 pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.46 to 1.04], Standard Error of Mean 0.64 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cognitive Remediation vs Active Control; Linear mixed effects model adjusted for age, sex, education (school years), comorbidities score (0-10), pain, Duke score (cardiac fitness), and cognitive status (MCI or cognitively normal) were used to compare changes in the mental health score of the SF-12 pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-1.04 to 1.85], Standard Error of Mean 0.73 — [estimate comment as in outcome 1, analysis 1]

21. Other Pre Specified Outcome: Falls.
Description: Presence and number of falls over 12 months from baseline.
Time Frame: Baseline and 12 Months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Number of Participants With Progression in Cognitive Impairment From Normal Cognitive Function at Baseline to Mild Cognitive Impairment (MCI)
Description: Progression in cognitive impairment from normal cognitive function at baseline to MCI.
Time Frame: Baseline and 2 Months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Number of Participants With Progression in Cognitive Impairment From Normal Cognitive Function at Baseline to Dementia
Description: Progression in cognitive impairment from baseline normal cognitive function to dementia.
Time Frame: Baseline and 2 Months
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Number of Participants With Progression in Cognitive Impairment From Normal Cognitive Function at Baseline to Motoric Cognitive Risk Syndrome (MCR)
Description: Progression in cognitive impairment from baseline normal cognitive function to MCR.
Time Frame: Baseline and 2 Months
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Number of Participants With Progression in Cognitive Impairment From Normal Cognitive Function at Baseline to Cognitively Impaired
Description: Progression in cognitive impairment from baseline normal cognitive function to cognitive impairment defined as presence of incident MCI, dementia, or MCR.
Time Frame: Baseline and 2 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months from intervention
Description: Participants were asked if they had any falls or changes in their health at bimonthly phone calls between study visits
Arm/Group | Cognitive Remediation | Active Control
All-Cause Mortality (participants affected / at risk) | 2/192 | 2/191
Serious Adverse Events (participants affected / at risk) | 5/192 | 1/191
Other Adverse Events (participants affected / at risk) | 49/192 | 34/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Remediation (N=192) | Active Control (N=191)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0)
High blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Remediation (N=192) | Active Control (N=191)
Fall (Musculoskeletal and connective tissue disorders) | 34 (41) | 34 (43)
Leg pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT02567227/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT02567227/ICF_001.pdf